CLINICAL TRIAL: NCT03440840
Title: Computer Training and Transcranial Direct Current Stimulation for Cognition in HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Raymond Ownby, M.D., Professor and Chair, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG056256
Record Dates: First submitted 2017-11-08; First posted 2018-02-22 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-11

CONDITIONS: HIV-related Mild Neurocognitive Disorder
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Cognitive Training

STUDY DESIGN:
Intervention Model Description: Randomized parallel group
Who Masked: Participant, Outcomes Assessor
Masking Description: Individuals will receive either active or sham tDCS. The outcomes assessor will be blind to treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Computer Training with active tDCS (Experimental): Participants randomized to this arm will receive computer-based cognitive training using a car racing game with active transcranial direct current stimulation (tDCS).
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS); Behavioral: Computer-based Cognitive Training
- Computer Training with sham tDCS (Active Comparator): Participants randomized to this arm will receive computer-based cognitive training using a car racing game with sham transcranial direct current stimulation (tDCS).
  Interventions: Behavioral: Computer-based Cognitive Training
- Computer Training with or without tDCS (Placebo Comparator): Participants in this arm will watch educational videos as a comparator to computer training with the car racing game (watching educational videos).
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS); Behavioral: Watching Educational Videos

INTERVENTIONS:
Procedure: Transcranial Direct Current Stimulation (tDCS) — Application of a small electrical current (1-2 mA) across the head.
  Other Names: tDCS
  Arms: Computer Training with active tDCS; Computer Training with or without tDCS
Behavioral: Computer-based Cognitive Training — Use of computer-delivered games or exercises with the goal of improving cognitive performance.
  Other Names: Cognitive Training
  Arms: Computer Training with active tDCS; Computer Training with sham tDCS
Behavioral: Watching Educational Videos — Watching educational videos and answering questions about them
  Arms: Computer Training with or without tDCS

SUMMARY:
This study investigates the effectiveness of computer-based cognitive training with or without transcranial direct current stimulation (tDCS) in improving the functioning of older individuals with HIV-related cognitive dysfunction.

DETAILED DESCRIPTION:
In spite of advances in its treatment, persons with HIV continue to develop HIV-associated neurocognitive disorders (HAND) over time. HAND may be an even more significant problem in older persons (age 50+) with HIV who may experience age-related changes in cognition in addition to HAND. Because of HAND's impact on patients' functioning and quality of life, treatments are needed. Pharmacologic treatments have, in general, been ineffective and investigators have argued that computer delivered cognitive training may be an effective alternative. While results of small studies have been encouraging, the effect size of cognitive training may be small and of unclear practical importance. The nature of cognitive training programs, often building on laboratory measures of cognition, may reduce how inherently interesting (i.e., fun) they are, limiting their uptake outside of paid research studies. Others have argued for the use of computer games targeting psychomotor speed, problem solving, and visuospatial skills to improve cognitive function in older adults. Data support the utility of this approach, but again effect sizes may be small.

Transcranial direct current stimulation (tDCS) may be an effective way to enhance the effects of cognitive training. It involves the application of a small electric current (1-2 mA) to the head, inducing small currents within the brain that enhance cognitive training. Multiple studies have shown that tDCS enhances cognition, including attention and psychomotor speed. The investigators previously completed a single-blind pilot study of individuals with HIV-related mild neurocognitive disorder using a high-interest car racing game with or without tDCS. Results were encouraging in showing moderate to large effect sizes consistent with tDCS enhancement of cognitive function after six 20-minute training sessions over two weeks. Participants' subjective reports of cognitive difficulties supported observed effects on objective measures, and their mood improved. The intervention was acceptable to participants, many of whom stated they enjoyed it. Everyone indicated a willingness to participate in a similar study in the future.

In this study the investigators will expand on a pilot-tested training intervention with 120 individuals randomly assigned to an attention control condition or game-based cognitive training with either sham or active tDCS. The investigators will employ a battery of cognitive measures as well as self-report measures of mood, cognitive difficulties, and everyday functioning in order to evaluate the effects of study interventions.

Participants will first be screened for eligibility by telephone, and then scheduled for a visit during which their eligibility will be further assessed. Those who are eligible based on inclusion and exclusion criteria will complete a battery of measures of their cognitive and functional status. They will then complete six training sessions over a period of three weeks, and then once again complete the battery of assessments. Participants will then be asked to return one month after the post-training assessment to evaluate the persistence of training effects.

ELIGIBILITY:
Inclusion Criteria:

* Treated with antiretroviral medication for at least one month
* Meet criteria for Mild Neurocognitive Disorder

Exclusion Criteria:

* Seizure disorder
* Recent head injury or surgery
* Personal or family history of bipolar disorder;
* Some medications
* Left handedness
* HIV Dementia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond L Ownby, MD, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- NSU Psychiatry Research Office, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
After the conclusion of the study, de-identified study data will be shared by the study principal investigator with interested individuals.
Supporting Information: Study Protocol
Time Frame: After study conclusion.
Access Criteria: Researchers who indicate an interest in using the data for legitimate purposes.

REFERENCES:
- [Background] Ownby RL, Acevedo A. A pilot study of cognitive training with and without transcranial direct current stimulation to improve cognition in older persons with HIV-related cognitive impairment. Neuropsychiatr Dis Treat. 2016 Oct 25;12:2745-2754. doi: 10.2147/NDT.S120282. eCollection 2016. PMID 27822047
- [Result] Ownby RL, Kim J. Computer-Delivered Cognitive Training and Transcranial Direct Current Stimulation in Patients With HIV-Associated Neurocognitive Disorder: A Randomized Trial. Front Aging Neurosci. 2021 Nov 15;13:766311. doi: 10.3389/fnagi.2021.766311. eCollection 2021. PMID 34867291

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Computer Training With Active tDCS | Computer Training With Sham tDCS | Computer Training With or Without tDCS
Started | 16 | 15 | 15
Completed | 15 | 14 | 15
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Computer Training With Active tDCS | Computer Training With Sham tDCS | Computer Training With or Without tDCS | Total
Number analyzed (Participants) | 16 | 15 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.06 (4.99) | 58.80 (4.13) | 61.07 (6.29) | 58.93 (5.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 9
  Male | 13 | 13 | 11 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 0 | 6
  Not Hispanic or Latino | 13 | 12 | 15 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 8 | 10 | 29
  White | 5 | 7 | 5 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 15 | 46
Psychomotor Speed [Mean (Standard Deviation); unit: units on a scale] — The Coding subtest of the Wechsler Adult Intelligence Scale, 4th ed. (WAIS-IV) asks that the person assessed insert small geometric drawings with pencil on paper according to a key at the top of the page. One figure corresponds to the numeral 1, another to 2, and so on. The persons is asked to work as quickly as they can, and given a specific period in which to complete the task. Raw scores are the number of boxes correctly filled in during the time allowed and can range from 0 to 155, with higher scores indicating a better performance.
  units on a scale | 48.94 (9.28) | 51.67 (13.70) | 46.07 (15.52) | 48.89 (12.93)
Functional Status [Mean (Standard Deviation); unit: units on a scale] — The University of California--San Diego Performance Based Skills Assessment, version B. The person assessed is asked to complete several functional tasks, including pretending to make a call on a telephone to change a medical appointment and paying an electric bill by filling out a check. Scores on the first task range form 0 to 9, and from 0 to 11 on the second. These raw scores are then converted to create a final combined score that ranges from 0 to 100, with higher scores indicating a better performance.
  units on a scale | 79.75 (10.71) | 80.20 (19.39) | 76.73 (13.72) | 78.91 (13.52)
Participant Assessment of Own Functioning (PAOF) [Mean (Standard Deviation); unit: units on a scale] — Participant self-report of problems related to cognitive and sensory functioning on the Participant Assessment of Own Functioning (PAOF). The PAOF includes 33 items ranged from 0 to 5, allowing a total score from 0 to 165. A higher score on this measure means that the person is reporting greater frequency with some mental activities.
  units on a scale | 8.18 (2.34) | 7.65 (4.46) | 8.55 (2.49) | 8.13 (2.40)
Center for Epidemiological Studies Depression Scale (CES-D) [Mean (Standard Deviation); unit: units on a scale] — Participant self-report of mood. The Center for Epidemiological Studies Depression scale (CES-D) is a self-report measure of symptoms of and related to depressed mood. It includes 20 items that are scored from 0 to 3 and summed for an overall score ranging from 0 to 60. Higher scores on this measure indicate that the person assessed is reporting a greater frequency or severity of depressive symptoms.
  units on a scale | 14.00 (7.55) | 15.27 (9.24) | 15.13 (7.19) | 14.78 (7.87)

OUTCOME MEASURES:

1. Primary Outcome: Psychomotor Speed
Description: Ability of the participant to attend to and use complex stimuli while making a motor response. The Coding subtest of the Wechsler Adult Intelligence Scale, 4th ed. (WAIS-IV) asks that the person assessed insert small geometric drawings with pencil on paper according to a key at the top of the page. One figure corresponds to the numeral 1, another to 2, and so on. The persons is asked to work as quickly as they can, and given a specific period in which to complete the task. Raw scores are the number of boxes correctly filled in during the time allowed and can range from 0 to 155, with higher scores indicating a better performance.
Time Frame: 3 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Computer Training With Active tDCS | Computer Training With Sham tDCS | Computer Training With or Without tDCS
Number analyzed (Participants) | 15 | 14 | 15
score on a scale | 54.2 [43.2 to 65.2] | 60.4 [49.4 to 71.4] | 53.4 [42.6 to 64.2]
Statistical Analysis 1: Comparison: Computer Training With Active tDCS vs Computer Training With or Without tDCS; Test type: Superiority; p = 0.40, Mixed Models Analysis; Estimated marginal means comparisons, Tukey adjustment; Mean Difference (Final Values) = 2.29, Standard Error of Mean 2.68

2. Secondary Outcome: Functional Status
Description: Participant performance on observed tasks of daily living. Participants completed the University of California--San Diego Performance Based Skills Assessment, version B. The person assessed is asked to complete several functional tasks, including pretending to make a call on a telephone to change a medical appointment and paying an electric bill by filling out a check. Scores on the first task range form 0 to 9, and from 0 to 11 on the second. These raw scores are then converted to create a final combined score that ranges from 0 to 100, with higher scores indicating a better performance.
Time Frame: 3 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Computer Training With Active tDCS | Computer Training With Sham tDCS | Computer Training With or Without tDCS
Number analyzed (Participants) | 15 | 14 | 15
score on a scale | 84.6 [74.8 to 94.5] | 82.8 [72.9 to 92.6] | 84.4 [74.8 to 94.0]
Statistical Analysis 1: Comparison: Computer Training With Active tDCS vs Computer Training With or Without tDCS; Test type: Superiority; p = 0.37, Mixed Models Analysis — Estimated marginal means comparisons, Tukey adjustment; Mean Difference (Final Values) = 1.86, Standard Error of Mean 2.04

3. Secondary Outcome: Participant Assessment of Own Functioning (PAOF)
Description: Participant self-report of problems related to cognitive and sensory functioning on the Participant Assessment of Own Functioning (PAOF). This is a self-report measure of the frequency with which a person experiences difficulties with various mental and sensory tasks, such as remembering what is said to them, understanding or expressing themselves in language, and thinking about complex problems. The PAOF includes 33 items ranged from 0 to 5, allowing a total score from 0 to 165. A higher score on this measure means that the person is reporting greater frequency with some mental activities.
Time Frame: 3 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Computer Training With Active tDCS | Computer Training With Sham tDCS | Computer Training With or Without tDCS
Number analyzed (Participants) | 15 | 14 | 15
score on a scale | 7.98 [6.27 to 9.69] | 7.73 [6.01 to 9.44] | 7.86 [6.19 to 9.52]
Statistical Analysis 1: Comparison: Computer Training With Active tDCS vs Computer Training With or Without tDCS; Test type: Superiority; p = 0.37, Mixed Models Analysis; Comparison of estimated marginal means, Tukey adjustment for multiple comparisons; Mean Difference (Final Values) = 1.86, Standard Error of Mean 2.04

4. Secondary Outcome: Center for Epidemiological Studies Depression Scale (CES-D)
Description: Participant self-report of mood. The Center for Epidemiological Studies Depression scale (CES-D) is a self-report measure of symptoms of and related to depressed mood. It includes 20 items that are scored from 0 to 3 and summed for an overall score ranging from 0 to 60. Higher scores on this measure indicate that the person assessed is reporting a greater frequency or severity of depressive symptoms.
Time Frame: 3 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Computer Training With Active tDCS | Computer Training With Sham tDCS | Computer Training With or Without tDCS
Number analyzed (Participants) | 15 | 14 | 15
score on a scale | 16.5 [9.53 to 23.50] | 16.6 [9.59 to 23.70] | 16.3 [9.54 to 23.10]
Statistical Analysis 1: Comparison: Computer Training With Active tDCS vs Computer Training With or Without tDCS; Test type: Superiority; p = 0.61, Mixed Models Analysis; Mean Difference (Final Values) = 1.42, Standard Error of Mean 2.77 — Differences between estimated marginal means, Tukey correction for multiple comparisons

ADVERSE EVENTS:
Time Frame: 7 weeks
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Computer Training With Active tDCS | Computer Training With Sham tDCS | Computer Training With or Without tDCS
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/16 | 1/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Computer Training With Active tDCS (N=16) | Computer Training With Sham tDCS (N=15) | Computer Training With or Without tDCS (N=15)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Reactivation of traumatic memories (Nervous system disorders) | 1 (1) | 0 (0) | 0

LIMITATIONS AND CAVEATS:
In this trial, we were only able to recruit 46 participants, of whom 44 completed the study. The original plan was to recruit 120 individuals, of whom 90 would complete the study. The sample size is thus substantially smaller than planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT03440840/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT03440840/SAP_001.pdf